CLINICAL TRIAL: NCT04080869
Title: Formulation of Retinyl Palmitate-loaded Topical Ethosomes for Treatment of Acne Vulgaris: a Split-face Comparative Clinical Study
Brief Title: Retinyl Palmitate-loaded Ethosomes in Acne Vulgaris
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sara Mohamed Awad, Assistant Professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RP-AV
Record Dates: First submitted 2019-09-04; First posted 2019-09-06 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Facial Acne Vulgaris
Keywords: acne vulgaris; retinoids; retinyl palmitate; ethosomes
MeSH Terms: conditions — Acne Vulgaris | interventions — retinol palmitate; Tretinoin

STUDY DESIGN:
Intervention Model Description: A Prospective, split face comparative clinical study
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The topical preparations are packed in non-identifiable jars and coded by a person who is not involved in the study the patient.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- retinyl palmitate ethosomes arm (Experimental): All patients will be instructed to apply a thin film of the new formula on one side of the face
  Interventions: Drug: retinyl palmitate
- tretinoin arm (Active Comparator): All patients will be instructed to apply a thin film of topical retinoid cream on the other side of the face
  Interventions: Drug: Tretinoin

INTERVENTIONS:
Drug: retinyl palmitate — topical retinyl palmitate loaded ethosomes
  Other Names: retinyl palmitate ethosomes
  Arms: retinyl palmitate ethosomes arm
Drug: Tretinoin — topical tretinoin
  Other Names: classic retinoid
  Arms: tretinoin arm

SUMMARY:
Acne is a chronic inflammatory dermatosis of the pilosebaceous unit. Topical treatment is the first choice in mild and moderate cases of acne, especially topical retinoids. Although topical retinoids are very effective in the treatment of acne, local cutaneous irritation including burning, itching, erythema, peeling or dryness, is observed in a considerable number of patients, resulting in low patient compliance, compromising the efficacy of the therapy.

Several approaches have been proposed to address these concerns, including the use of esters of retinoic acid (RA) and RA precursors, such as retinol and retinaldehyde, or novel drug delivery systems, which present the potential for controlled release, in turn reducing the aforementioned occurrences.

Encapsulation of retinoids into vesicular carriers as liposomes and ethosomes and nanoparticulate carriers can significantly improve their effects for the treatment of acne compared with commercial formulations , providing better tolerability of irritating retinoid.

The aim of work is to assess the efficacy and tolerability of the topical application of Retinyl Palmitate-loaded ethosome formulation in the treatment of acne vulgaris in comparison to conventional formulation of classic retinoids

ELIGIBILITY:
Inclusion Criteria:

* Patients with facial mild to moderate acne vulgaris
* Patients aged 12-40 years old

Exclusion Criteria:

* Pregnant females
* Patients with skin condition of the face such as rosacea, perioral dermatitis, atopic or seborrheic dermatitis or psoriasis.
* Patients with known hypersensitivity to preparations containing retinoid.
* Patients who take any other cocomitant systemic or topical medications for acne vulgaris

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2020-08-28 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Efficacy of the medication: number of inflammatory, non-inflammatory and total lesions | at first and every 2 weeks during the 6-week treatment period from starting the topical application
  counting the number of inflammatory, non-inflammatory and total lesions at first and every week during the treatment
assessment of tolerability: interviewing the patients | every 2 weeks during the 6-week treatment period from starting the topical application
  interviewing the patients about any sign/symptom of adverse reactions (erythema, peeling, burning sensation, dryness and pruritus)

CONTACTS AND LOCATIONS:
Overall Officials: Sara M Awad, MD, Principal Investigator — Department of Dermatology, Venereology and Andrology, Assiut University Hospital
Locations (1):
- Assiut University Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes
data that underlie results in a publication
Supporting Information: Study Protocol, SAP, CSR
Time Frame: starting 6 months after publication

REFERENCES:
- [Background] Manconi M, Valenti D, Sinico C, Lai F, Loy G, Fadda AM. Niosomes as carriers for tretinoin. II. Influence of vesicular incorporation on tretinoin photostability. Int J Pharm. 2003 Jul 24;260(2):261-72. doi: 10.1016/s0378-5173(03)00268-0. PMID 12842345
- [Result] Castro GA, Ferreira LA. Novel vesicular and particulate drug delivery systems for topical treatment of acne. Expert Opin Drug Deliv. 2008 Jun;5(6):665-79. doi: 10.1517/17425247.5.6.665. PMID 18532922
- [Result] Date AA, Naik B, Nagarsenker MS. Novel drug delivery systems: potential in improving topical delivery of antiacne agents. Skin Pharmacol Physiol. 2006;19(1):2-16. doi: 10.1159/000089138. PMID 16247244